CLINICAL TRIAL: NCT02171702
Title: A Phase I Open Label Dose Escalation Study of Once-daily Oral Treatment With BIBW 2992 for 28 Days in Patients With Advanced Solid Tumours
Brief Title: Dose Escalation Study of Oral Treatment With BIBW 2992 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.3
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (3):
- BIBW 2992 (Experimental): dose escalation
  Interventions: Drug: BIBW 2992
- BIBW 2992, fasted (Experimental): food effect part: maximum tolerated dose of BIBW 2992
  Interventions: Drug: BIBW 2992
- BIBW 2992, fed (Experimental): food effect part: maximum tolerated dose of BIBW 2992
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992

SUMMARY:
The primary objective of the study was to identify the maximum tolerated dose and to evaluate safety, pharmacokinetics, pharmacodynamic parameters, and efficacy of BIBW 2992.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of advanced, non-resectable and / or metastatic solid tumours, of types historically known to express EGFR and/or HER2, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment preferably patients with breast, colorectal or prostate cancer
* Age 18 years or older
* Life expectancy of at least three (3) months
* Written informed consent that is consistent with International Conference on Harmonization - Good Clinical Practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2
* Patients completely recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies to CTC <= Grade 1
* Patients must be recovered from previous surgery

The 12 additional patients recruited at the MTD must also meet the following criteria:

* Measurable tumour deposits (RECIST) by one or more techniques (X-ray, CT, MRI) and/or recognized tumour markers such as prostate-specific antigen prostate cancer) or cancer antigen 125 (Ovarian cancer)

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least eight (8) weeks, no history of cerebral edema or bleeding in the past eight (8) weeks and no requirement for steroids or anti-epileptic therapy
* Cardiac left ventricular function with resting ejection fraction CTC >= Grade 1
* Absolute neutrophil count (ANC) less than 1500 / mm3
* Platelet count less than 100 000 / mm3
* Bilirubin greater than 1.5 mg /dl (>26 μmol /L, Système Internationale (SI) unit equivalent)
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg / dl (>132 μmol / L, SI unit equivalent)
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast-feeding
* Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (excluding Luteinizing Hormone-Releasing Hormone agonists, or other hormones taken for breast cancer, or bisphosphonates), or participation in another clinical study within the past 4 weeks before start of therapy or concomitantly with this study
* Treatment with an EGFR- or HER2 inhibiting drug within the past four weeks before start of therapy or concomitantly with this study (8 weeks for trastuzumab)
* Patients unable to comply with the protocol
* Active alcohol or drug abuse

A patient may be eligible for re-treatment after the previous course is finished. A patient will not be eligible if any of the following conditions are met.

* Patients with clinical signs of disease progression or if latest X-ray, CT or MRI reveals Progressive Disease
* Cardiac left ventricular function CTC >= Grade 2 at any time during the previous course
* Patients fulfilling any of the Exclusion Criteria listed before as determined before treatment on Day 28, R5 of the previous course
* Patient not recovered from any dose-limiting toxicity 14 days after the last administration of BIBW 2992 in the previous course. Recovery is defined as return to baseline level or CTC Grade 1, whichever is higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-11; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of BIBW 2992 | up to 24 weeks
Incidence and intensity of Adverse Events according to Common Toxicity Criteria (CTC version 3) associated with increasing doses of BIBW 2992 | up to 28 weeks

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) for several time points | up to 648 hours after first drug administration, pre-dose on day 15 and 28
Percentage of AUC0-∞ that is obtained by extrapolation (%AUCtz-∞) | up to 648 hours after first drug administration, pre-dose on day 15 and 28
predose plasma concentration | predose on days 8, 15, 22 and 27
Plasma concentration | 24 hours after drug administration on the first (C24,1) and the Day 27 dose (C24,27)
Maximum measured plasma concentration (Cmax) for several time points | up to 648 hours after first drug administration, pre-dose on day 15 and 28
Time from dosing to the maximum plasma concentration (tmax) for several time points | up to 648 hours after first drug administration, pre-dose on day 15 and 28
terminal half-life (t1/2(ss)) | up to 648 hours after first drug administration, pre-dose on day 15 and 28
mean residence time after oral administration (MRTpo(ss)) | up to 648 hours after first drug administration, pre-dose on day 15 and 28
apparent clearance (CL/F(ss)) | up to 648 hours after first drug administration, pre-dose on day 15 and 28
apparent volume of distribution during the terminal phase (Vz/F(ss)) | up to 648 hours after first drug administration, pre-dose on day 15 and 28
Accumulation ratio between Day 1 and Day 27 with respect to Cmax (RA1) and AUC (RA2) | up to 648 hours after first drug administration, pre-dose on day 15 and 28
Modulation of biomarker (EGFR, p-EGFR, p-MAPK, p-Akt, Ki 67, p-27KIP1) in skin biopsies | Baseline and day 28 of the first treatment period
Modulation of biomarker (EGFR, p-EGFR, HER2 (Class I Tyrosine Kinase Receptor), p-MAPK (mitogen-activated protein kinase), p-Akt, Ki 67, p-27KIP1) in tumour biopsies in six or more patients treated at the MTD | Baseline and day 28 of the first treatment period
Objective tumour response | up to 25 weeks
Correlation of EGFR, HER2, estrogen receptor (ER) and progesterone receptor (PrR) immunohistochemical status as based on tumour biopsies, or excisions obtained prior to this study, with objective tumour responses | up to 25 weeks